CLINICAL TRIAL: NCT03189797
Title: Effect of Tailored Preventive Program on Caires Incidence Using International Caries Classification and Management System (ICCMS) A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mamdouh, Internal resident at operative department cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEBC-CU-2017-03-15
Record Dates: First submitted 2017-06-12; First posted 2017-06-16 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: A total number of 144 high caries risk dental students are selected based on the applied caries risk assessment method (CAMBRA). In the study group they are given a preventive program as homecare program including tooth brushing 2/day with a fluoride toothpaste( 5000 ppm F) in addition to fluoride mouth rinse. For the clinical approach motivational engagement isdone by discussing with patients how to improve oral health behavior including amount of sugar, fibrous food and junk food. This in addition to pits and fissures sealant, F- varnish 2 times /year.application of fluoride varnish every 6 months and dietary intake interventions.
  In the Control group participants assigned to the control condition will be advised to maintain their existing lifestyles. For ethical reasons, if the program shows its effectiveness, it will be made available to all groups at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): After defining the individual patient's likelihood risk status and the diagnosis for each lesion, ICCMS presents a management element to build a comprehensive patient care plan as follow:
  In the study group they were given a preventive program as homecare program including tooth brushing 2/day with a fluoride toothpaste( 5000 ppm F) following the instructions in addition to fluoride mouth rinse. For the clinical approach motivational engagement was done by discussing with patients how to improve oral health behavior including amount of sugar, fibrous food and junk food. This in addition to pits and fissures sealant, F- varnish 2 times /year. and application of fluoride varnish every 6 months and dietary intake interventions.
  Interventions: Other: tailored preventive program
- control group (No Intervention): In the Control group participants assigned to the control condition will be advised to maintain their existing lifestyles. For ethical reasons, if the program shows its effectiveness, it will be made available to all groups at the end of the study.

INTERVENTIONS:
Other: tailored preventive program — In the study group they were given a preventive program as homecare program including tooth brushing 2/day with a fluoride toothpaste( 5000 ppm F) following the instructions in addition to fluoride mouth rinse. For the clinical approach motivational engagement was done by discussing with patients how to improve oral health behavior including amount of sugar, fibrous food and junk food. This in addition to pits and fissures sealant, F- varnish 2 times /year. and application of fluoride varnish every 6 months and dietary intake interventions.
  Other Names: preventive dental program
  Arms: study group

SUMMARY:
This study will be conducted to evaluate The Effect of tailored preventive program on caries incidence using International Caries Classification and Management System (ICCMS) at a follow up periods of 3 ,6 and 12 months.

DETAILED DESCRIPTION:
A total number of 144 high caries risk dental students were selected based on the applied caries risk assessment method (CAMBRA). In the study group they were given a preventive program as homecare program including tooth brushing 2/day with a fluoride toothpaste( 5000 ppm F) following the instructions in addition to fluoride mouth rinse. For the clinical approach motivational engagement was done by discussing with patients how to improve oral health behavior including amount of sugar, fibrous food and junk food. This in addition to pits and fissures sealant, F- varnish 2 times /year. Recalls up were done at 3, 6 and 12 months by recording the caries prevalence , application of fluoride varnish every 6 months and dietary intake interventions. In the Control group participants assigned to the control condition will be advised to maintain their existing lifestyles. For ethical reasons, if the program shows its effectiveness, it will be made available to all groups at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Dental student.
* No malocclusion.
* Medically free

Exclusion Criteria:

* Compromised medical history.
* Severe or active periodontal disease.
* Heavy bruxism or a traumatic occlusion

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of dental caires | baseline
  ICCMS caries index
  Before the dental educational program, an oral examination will be done for the patient. Examination will be done by using mouth mirror and probe in natural day light. The educational program and outcome assessment will be assessed by ICCMS three times (immediately, three and six months) as the follow:
  Score 0 Tooth surfaces show no evidence of visible caries (no or questionable change in enamel translucency). Score 1 First or distinct visual changes in enamel seen as a carious opacity or visible discolouration not consistent with clinical appearance of sound enamel and which show no evidence of surface breakdown or underlying dentine shadowing.
  Score 2 A white or brown spot lesion with Localised enamel breakdown, without visible dentine exposure.
  Extensive stage Score 3 A distinct cavity in opaque or discoloured enamel with visible dentine.
Incidence of dental caires | 3 months
  ICCMS caries index
Incidence of dental caires | 6 months
  ICCMS caries index
Incidence of dental caires | 12 months
  ICCMS caries index

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mamdouh, Cairo, Maadi, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garcia RI, Sohn W. The paradigm shift to prevention and its relationship to dental education. J Dent Educ. 2012 Jan;76(1):36-45. PMID 22262548
- Available data/document: Study Protocol — https://www.ncbi.nlm.nih.gov/pubmed